CLINICAL TRIAL: NCT01557101
Title: Effectiveness of Colon Capsule Endoscopy as Colorectal Cancer Method of Screening in The Familiar-Risk Population
Brief Title: Comparison Colon Capsule Endoscopy vs Optical Colonoscopy for Colorectal Cancer Screening in Familiar-Risk Population
Acronym: CRIBADO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEC_cribado_CCR
Record Dates: First submitted 2012-03-13; First posted 2012-03-19 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Cancer, Genetics of
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COLON CAPSULE ENDOSCOPY (Other)
  Interventions: Procedure: COLON CAPSULE ENDOSCOPY ADHERENCE
- OPTICAL COLONOSCOPY (Other)
  Interventions: Procedure: OPTICAL COLONOSCOPY ADHERENCE

INTERVENTIONS:
Procedure: COLON CAPSULE ENDOSCOPY ADHERENCE — An exploration with a COLON CAPSULE ENDOSCOPY eaten which capsule has a video-camera in both end to see the colon.
  Arms: COLON CAPSULE ENDOSCOPY
Procedure: OPTICAL COLONOSCOPY ADHERENCE — An exploration with an OPTICAL COLONOSCOPY from the anus to see the colon.
  Arms: OPTICAL COLONOSCOPY

SUMMARY:
The purpose of this study is to determine if the adherence to screening in first grade relatives of patients with CCR is higher than optical colonoscopy.

DETAILED DESCRIPTION:
The purpose of this study is to compare the adherence and effectiveness of colon capsule endoscopy (CCE-2) versus conventional colonoscopy to screen first-degree relatives of patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic first-degree relatives (parents, siblings or children) of CRC patients aged less than 60 years or with two or more first-degree relatives of any age.
* Signing of informed consent.

Exclusion Criteria:

* Personal history of adenoma or CRC.
* History of hereditary CRC.
* Chronic inflammatory disease.
* Presence of digestive symptoms.
* Patients with swallowing problems (dysphagia).
* Personal history of gastrointestinal surgery.
* Enteritis radioactive.
* Renal failure.
* Congestive heart failure
* Allergy or other contraindication to Bysacodyl to PEG or phosphates.
* Pregnancy.
* Suspected bowel obstruction or intestinal strictures or fistulas known.
* Colectomy.
* Paralysis with impaired intestinal motility.
* Any other process that the investigator's discretion to make inadequate participation.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Participation to colorectal cancer screening in first-degree relatives of patients with colorectal cancer | 6 month follow up
  Assess whether colon capsule endoscopy increases participation to colorectal cancer screening in first-degree relatives of patients with colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Quintero, MD. PhD., Principal Investigator — Hospital Universitario de Canarias
Locations (2):
- Spain (2):
  - Digestive Service, Huc, San Cristóbal de La Laguna, S/c de Tenerife
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, S/c de Tenerife

REFERENCES:
- [Derived] Adrian-de-Ganzo Z, Alarcon-Fernandez O, Ramos L, Gimeno-Garcia A, Alonso-Abreu I, Carrillo M, Quintero E. Uptake of Colon Capsule Endoscopy vs Colonoscopy for Screening Relatives of Patients With Colorectal Cancer. Clin Gastroenterol Hepatol. 2015 Dec;13(13):2293-301.e1. doi: 10.1016/j.cgh.2015.06.032. Epub 2015 Jun 29. PMID 26133904